CLINICAL TRIAL: NCT04856865
Title: A Phase 1/2, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of ADP101 for Oral Immunotherapy in Food-Allergic Children and Adults (The Harmony Study)
Brief Title: ADP101 for Oral Immunotherapy in Food-Allergic Children and Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alladapt Immunotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADP101-MA-01
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Food Allergy
Keywords: ADP101; Allergy; Oral immunotherapy; OIT; Allergies; Food allergies; Multi-food allergic; Multi-allergen oral immunotherapy; Tree nut allergy; Milk allergy; Wheat allergy; Egg allergy; Fin fish allergy; Shrimp allergy; Peanut allergy; Sesame seed allergy; Soy allergy; Shellfish allergy; Fish allergy; Seafood allergy; Dairy allergy; Desensitization; Food hypersensitivity; Immune system disease; Hypersensitivity, immediate; Hypersensitivity
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity; Nut Hypersensitivity; Milk Hypersensitivity; Wheat Hypersensitivity; Egg Hypersensitivity; Peanut Hypersensitivity; Shellfish Hypersensitivity; Immune System Diseases; Hypersensitivity, Immediate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose ADP101 (Experimental): Participants received ADP101 at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 1500mg ADP101 over the 40 week treatment period. ADP101: Oral formulation mixture of 15 individual food sources from commercially available food flours containing allergenic proteins (almond, cashew, chicken's egg, codfish, cow's milk, hazelnut, peanut, pecan, pistachio, salmon, sesame seed, shrimp, soy, walnut, and wheat) with excipients. Each dose is formulated to contain equal parts by protein weight of each of the 15 individual foods in ADP101.
  Interventions: Biological: Low dose ADP101
- High dose ADP101 (Experimental): Participants received ADP101 at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 4500mg ADP101 over the 40 week treatment period. ADP101: Oral formulation mixture of 15 individual food sources from commercially available food flours containing allergenic proteins (almond, cashew, chicken's egg, codfish, cow's milk, hazelnut, peanut, pecan, pistachio, salmon, sesame seed, shrimp, soy, walnut, and wheat) with excipients. Each dose is formulated to contain equal parts by protein weight of each of the 15 individual foods in ADP101.
  Interventions: Biological: High dose ADP101
- Pooled Placebo (Experimental): Participants received volume-matched placebo at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 1500mg or 4500mg placebo over the 40 week treatment period. Placebo: Powder containing excipient, aroma and flavor maskers, and coloring agents to achieve similar appearance and total weight as the active, in the same cup packaging as the active.
  Interventions: Biological: Pooled Placebo

INTERVENTIONS:
Biological: Low dose ADP101 — Active powder formulation
  Other Names: 1500mg target dose ADP101
  Arms: Low dose ADP101
Biological: High dose ADP101 — Active powder formulation.
  Other Names: 4500mg target dose ADP101
  Arms: High dose ADP101
Biological: Pooled Placebo — Placebo powder
  Other Names: Placebo
  Arms: Pooled Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ADP101 in food allergic children and adults.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study of the efficacy and safety of ADP101 for oral immunotherapy in food allergic children and adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 55 (inclusive)
* Clinical history of allergy to at least 1 of the foods contained in ADP101
* Experience dose-limiting symptoms at or below the 100-mg dose level to 1 or multiple food sources in ADP101

Exclusion Criteria:

* Experience dose limiting symptoms at or below the 100 mg challenge dose level to more than 5 food sources contained in ADP101
* History of severe or life-threatening episode(s) of anaphylaxis or anaphylactic shock within 60 days of screening
* History of EoE, other eosinophilic gastrointestinal disease, chronic, recurrent or severe GERD, symptoms of dysphagia
* Severe asthma
* Mild or moderate asthma, if uncontrolled or difficult to control
* History of mast cell disorder, including mastocytosis, urticaria pigmentosa or angioedema
* History of chronic disease (other than asthma, atopic dermatitis, or allergic rhinitis) at risk of becoming unstable or requiring a change in chronic therapeutic regimen e.g. uncontrolled diabetes
* History of cardiovascular disease, including hypertension requiring > 2 antihypertensive medications
* History of interstitial lung disease
* History of celiac disease
* Active autoimmune disease that has required systemic treatment within 3 months
* Known malignancy that is progressing or has required active treatment within the past 3 years
* Known history of HIV, known active hepatitis B infection or known active hepatitis C virus infection
* Prior/concurrent therapies as follows:

  * beta-blockers, ACE inhibitors, ARBs or calcium channel blockers
  * regular steroid medication use
  * therapeutic antibody treatment currently or within the previous 6 months
  * any food immunotherapy currently or within the previous 12 weeks
  * In the build up phase of non-food immunotherapy
* Residing at the same address as another subject (e.g. siblings) participating in this or any other OIT study
* Develops dose-limiting symptoms to placebo during the Screening DBPCFC
* Any other condition that might preclude safe participation in the study

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Lun Wang, MD, Study Director — VP of Clinical Development, Alladapt Immunotherapeutics, Inc.
Locations (15):
- United States (15):
  - Study Site, Mission Viejo, California
  - Study Site, Rolling Hills Estates, California
  - Study Site, San Diego, California
  - Study Site, Denver, Colorado
  - Study Site, Tampa, Florida
  - Study Site, Atlanta, Georgia
  - Study Site, Marietta, Georgia
  - Study Site, Normal, Illinois
  - Study Site, Ann Arbor, Michigan
  - Study Site, Chapel Hill, North Carolina
  - Study Site, Cincinnati, Ohio
  - Study Site, Happy Valley, Oregon
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Charleston, South Carolina
  - Study Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized in a 2:2:1:1 ratio to 1 of 4 arms, with 2 arms in each dosing regimen (low or high), to receive daily oral doses of study drug (either ADP101 or matching placebo) in a blinded fashion. Data from placebo participants (high-dose or low-dose) was analyzed in a pooled fashion (Pooled Placebo)
Period: Overall Study
Arm/Group | Low Dose ADP101 | High Dose ADP101 | Pooled Placebo
Started | 25 | 24 | 24
Completed | 19 | 16 | 21
Not Completed | 6 | 8 | 3

BASELINE CHARACTERISTICS:
Population: The ITT analysis is defined as all randomized participants, age 4-55 years
Groups:
- Pooled Placebo: Participants received volume-matched placebo at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 1500mg or 4500mg placebo (see randomization scheme in pre-assignment details) over the 40 week treatment period. Placebo: Powder containing excipient, aroma and flavor maskers, and coloring agents to achieve similar appearance and total weight as the active, in the same cup packaging as the active.
- Total: Total of all reporting groups
Arm/Group | Low Dose ADP101 | High Dose ADP101 | Pooled Placebo | Total
Number analyzed (Participants) | 25 | 24 | 24 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 20 | 20 | 61
  Between 18 and 65 years | 4 | 4 | 4 | 12
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (9.9) | 12.1 (6) | 14.8 (11.3) | 13.6 (9.3)
Age, Customized [Mean (Standard Deviation); unit: years] — The primary analysis population was the pediatric ITT population, age 4-17 years at the time of randomization Population: Primary analysis population was the pediatric ITT population, age 4-17 years at the time of randomization
  years
    Mean (SD) age (years) of pediatric ITT population: number analyzed (Participants) | 21 | 20 | 20 | 61
    Mean (SD) age (years) of pediatric ITT population | 10.3 (3.4) | 9.9 (2.8) | 10.1 (3.5) | 10.1 (3.2)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Primary analysis population was the pediatric ITT population, age 4-17 at the time of randomization
  Participants
    Gender: number analyzed (Participants) | 21 | 20 | 20 | 61
    Gender: Female | 7 | 6 | 7 | 20
    Gender: Male | 14 | 14 | 13 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 11 | 29
  Male | 15 | 16 | 13 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 0 | 5
  Not Hispanic or Latino | 23 | 20 | 22 | 65
  Unknown or Not Reported | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 2 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 3
  White | 18 | 20 | 14 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 24 | 73
Primary analysis population (pediatric ITT) [Count of Participants; unit: Participants] — The primary analysis population for the study was the pediatric ITT population, which included participants ages 4-17 years of age at the time of randomization.
  Participants | 21 | 20 | 20 | 61

OUTCOME MEASURES:

1. Primary Outcome: 600mg Desensitization in at Least One Qualifying Food
Description: The proportion of participants in the pediatric ITT population who tolerated the 600mg level of a single qualifying food without dose limiting symptoms at the Week 40 Exit DBPCFC.
Time Frame: 40 Weeks
Population: The primary analysis population was the pediatric ITT population, age 4-17 years at the time of randomization
Measure: Count of Participants; unit: Participants
Groups:
- Low Dose ADP101: Participants received ADP101 at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 1500mg ADP101 over the 40 week treatment period. ADP101:Oral formulation mixture of 15 individual food sources from commercially available food flours containing allergenic proteins (almond, cashew, chicken's egg, codfish, cow's milk, hazelnut, peanut, pecan, pistachio, salmon, sesame seed, shrimp, soy, walnut, and wheat) with excipients. Each dose is formulated to contain equal parts by protein weight of each of the 15 individual foods in ADP101.
- High Dose ADP101: Participants received ADP101 at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 4500mg ADP101 over the 40 week treatment period. ADP101:Oral formulation mixture of 15 individual food sources from commercially available food flours containing allergenic proteins (almond, cashew, chicken's egg, codfish, cow's milk, hazelnut, peanut, pecan, pistachio, salmon, sesame seed, shrimp, soy, walnut, and wheat) with excipients. Each dose is formulated to contain equal parts by protein weight of each of the 15 individual foods in ADP101.
- Pooled Placebo: Participants received volume-matched placebo at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 1500mg or 4500mg placebo over the 40 week treatment period. Placebo:Powder containing excipient, aroma and flavor maskers, and coloring agents to achieve similar appearance and total weight as the active, in the same cup packaging as the active.
Arm/Group | Low Dose ADP101 | High Dose ADP101 | Pooled Placebo
Number analyzed (Participants) | 21 | 20 | 20
Participants | 8 | 11 | 4

2. Secondary Outcome: 1000mg Desensitization Threshold in Pediatric ITT Population
Description: Proportion of participants in the pediatric ITT population (age 4-17 at randomization) who tolerated the 1000mg level of a single qualifying food without dose limiting symptoms at the Week 40 Exit DBPCFC.
Time Frame: 40 weeks
Population: Primary analysis population was the pediatric ITT population, age 4-17 years at the time of randomization
Measure: Count of Participants; unit: Participants
Groups:
- Pooled PBO: Participants received volume-matched placebo at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 1500mg or 4500mg placebo over the 40 week treatment period. Placebo:Powder containing excipient, aroma and flavor maskers, and coloring agents to achieve similar appearance and total weight as the active, in the same cup packaging as the active.
Arm/Group | Low Dose ADP101 | High Dose ADP101 | Pooled PBO
Number analyzed (Participants) | 21 | 20 | 20
Participants | 5 | 10 | 3

3. Secondary Outcome: 600mg Desensitization Threshold, Multi-allergic Pediatric ITT Population
Description: Proportion of participants with >=2 qualifying FAs in the pediatric ITT population (age 4-17 at randomization) who tolerated the 600mg level of each of 2 or more qualifying foods without dose limiting symptoms at the Week 40 Exit DBPCFC.
Time Frame: 40 weeks
Population: Primary analysis population is the pediatric ITT population age 4-17 years at the time of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose ADP101 | High Dose ADP101 | Pooled PBO
Number analyzed (Participants) | 21 | 20 | 20
Participants | 2 | 5 | 0

4. Secondary Outcome: 1000mg Desensitization Threshold, Multi-allergic Pediatric ITT Population
Description: Proportion of participants with >=2 qualifying FAs in the pediatric ITT population (age 4-17 at randomization) who tolerated the 1000mg level of each of 2 or more qualifying foods without dose limiting symptoms at the Week 40 Exit DBPCFC.
Time Frame: 40 Weeks
Population: The primary analysis population is the pediatric ITT population, age 4-17 years at the time of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose ADP101 | High Dose ADP101 | Pooled PBO
Number analyzed (Participants) | 21 | 20 | 20
Participants | 1 | 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from consent until 14 days after last dose of study drug, up to approximately 52 weeks of treatment. Serious adverse events (SAEs) considered related to ADP101 were to be reported at any time until resolution/stabilization of the SAE.
Description: Allergic reactions were graded according to the Consortium of Food Allergy Research (CoFAR grading system, Jones et al. 2017),including events that met the definition for anaphylaxis.
  The pediatric Safety population included all pediatric participants (age 4-17 at the time of randomization) who received at least one dose of study drug. The All-participants safety population included all participants (age 4-55 years at the time of randomization) who received at least one dose of study drug.
Groups:
- Low Dose ADP101, Pediatric Safety Population; Low Dose ADP101, All-participants Safety Population: Participants received ADP101 at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 1500mg ADP101 over the 40 week treatment period.
- High Dose ADP101, Pediatric Safety Population; High Dose ADP101, All-participants Safety Population: Participants received ADP101 at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 4500mg ADP101 over the 40 week treatment period.
- Pooled PBO, Pediatric Safety Population; Pooled PBO, All-participants Safety Population: Participants received volume-matched placebo at a starting dose of 5mg po daily, with supervised updosing in the clinic as tolerated every 2 weeks to a target dose of 1500mg or 4500mg placebo over the 40 week treatment period.
Arm/Group | Low Dose ADP101, Pediatric Safety Population | High Dose ADP101, Pediatric Safety Population | Pooled PBO, Pediatric Safety Population | Low Dose ADP101, All-participants Safety Population | High Dose ADP101, All-participants Safety Population | Pooled PBO, All-participants Safety Population
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/20 | 0/25 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/20 | 0/20 | 0/25 | 1/24 | 0/24
Other Adverse Events (participants affected / at risk) | 20/21 | 19/20 | 19/20 | 24/25 | 23/24 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose ADP101, Pediatric Safety Population (N=21) | High Dose ADP101, Pediatric Safety Population (N=20) | Pooled PBO, Pediatric Safety Population (N=20) | Low Dose ADP101, All-participants Safety Population (N=25) | High Dose ADP101, All-participants Safety Population (N=24) | Pooled PBO, All-participants Safety Population (N=24)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose ADP101, Pediatric Safety Population (N=21) | High Dose ADP101, Pediatric Safety Population (N=20) | Pooled PBO, Pediatric Safety Population (N=20) | Low Dose ADP101, All-participants Safety Population (N=25) | High Dose ADP101, All-participants Safety Population (N=24) | Pooled PBO, All-participants Safety Population (N=24)
Abdominal pain (Gastrointestinal disorders) | 10 | 6 | 6 | 11 | 6 | 8
Nausea (Gastrointestinal disorders) | 9 | 7 | 2 | 12 | 8 | 4
Oral pruritis (Gastrointestinal disorders) | 5 | 7 | 5 | 9 | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 4 | 7 | 4 | 5 | 9 | 6
Vomiting (Gastrointestinal disorders) | 6 | 5 | 4 | 7 | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 7 | 5 | 2 | 9
Paresthesia oral (Gastrointestinal disorders) | 8 | 2 | 2 | 8 | 2 | 5
Abdominal discomfort (Gastrointestinal disorders) | 5 | 4 | 1 | 5 | 6 | 2
Tongue pruritis (Gastrointestinal disorders) | 4 | 2 | 1 | 4 | 2 | 1
Lip swelling (Gastrointestinal disorders) | 3 | 2 | 1 | 3 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2
Lip erythema (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Lip pruritis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 2 | 8 | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 5 | 8 | 4 | 6
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 5 | 5 | 6 | 7
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 5 | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 4 | 1 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 2 | 3 | 2
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 2 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 2 | 3 | 1
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 1 | 1
Nasal pruritis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 2 | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 1
Throat clearing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 6 | 7 | 6 | 8 | 9 | 6
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 2 | 5 | 6 | 3
Viral infection (Infections and infestations) | 2 | 3 | 3 | 2 | 3 | 3
Gastroenteritis viral (Infections and infestations) | 3 | 2 | 2 | 3 | 2 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 4 | 2 | 1 | 4
Ear infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 1
Otitis media (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Laryngitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 6 | 7 | 9 | 7 | 7
Pruritis (Skin and subcutaneous tissue disorders) | 7 | 5 | 3 | 8 | 5 | 6
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 4 | 3 | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 3 | 1 | 3
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | 0 | 5
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 8 | 9 | 11 | 10 | 11 | 13
Hypersensitivity (Immune system disorders) | 1 | 1 | 1 | 1 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 2 | 0 | 0 | 2
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 1 | 3 | 5 | 1 | 4
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Chest discomfort (General disorders) | 2 | 1 | 1 | 3 | 2 | 1
Pyrexia (General disorders) | 1 | 0 | 2 | 1 | 0 | 3
Fatigue (General disorders) | 2 | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 1
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Swelling face (General disorders) | 0 | 1 | 0 | 0 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 1 | 2
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 1 | 1
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Eye pruritis (Eye disorders) | 2 | 0 | 3 | 2 | 0 | 3
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 2
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0 | 1 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 2 | 0
Ear pruritis (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 1 | 0 | 1 | 1 | 1
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 0 | 1 | 1 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT04856865/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT04856865/SAP_001.pdf